CLINICAL TRIAL: NCT02666430
Title: An Open-label, Randomized, Multi-center, Parallel-Group Clinical Trial Comparing the Efficacy and Safety of Mylan's Insulin Glargine With Lantus® in Type 1 Diabetes Mellitus Patients: An Extension Study
Brief Title: Extension Study to Assess Safety and Efficacy of Mylan's Insulin Glargine and Lantus® in Type 1 Diabetes Mellitus (T1DM) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYL-1501D-3003
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mylan's insulin glargine (Experimental): Patients will be administered either Mylan insulin glargine or Lantus® subcutaneously, once daily in combination with lispro and titrated based on blood glucose readings per standard of care for a total of thirty-six (36) weeks, split into three cycles of twelve (12) weeks each.
  Interventions: Drug: Mylan's insulin glargine
- Lantus® (Active Comparator): Patients will be administered either Mylan insulin glargine or Lantus® subcutaneously, once daily in combination with lispro and titrated based on blood glucose readings per standard of care for a total of thirty-six (36) weeks, split into three cycles of twelve (12) weeks each.
  Interventions: Drug: Lantus®

INTERVENTIONS:
Drug: Mylan's insulin glargine
  Arms: Mylan's insulin glargine
Drug: Lantus®
  Arms: Lantus®

SUMMARY:
The aim of this extension study is to assess the safety and efficacy of Mylan's insulin glargine and Lantus® in T1DM patients.

DETAILED DESCRIPTION:
This multi-center, open-label, randomized clinical extension study in patients with T1DM will assess safety and efficacy of Mylan's insulin glargine and Lantus®.

Patients with an established diagnosis of T1DM per American Diabetes Association 2014 criteria who were randomized to the Lantus® treatment arm of the Mylan Glargine 3001 study, and who have completed the 52-week treatment period on Lantus® will be eligible to be screened for the MYL-1501D-3003 study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have completed the 52-week treatment period (irrespective of their age at the completion of MYL-GAI-3001 trial) of the MYL-GAI-3001 trial and were assigned to Lantus® in that study.
2. Patients or their legal representatives must give written and signed informed consent before starting any protocol-specific procedures.
3. The patient is able and willing to comply with the requirements of the extension study protocol including the 8-point self-monitoring blood glucose, completion of patient diary records as instructed and following a recommended diet and exercise plan for the entire duration of the extension study.
4. Female patients complying with the following:

   * Female patients of childbearing potential must be using oral contraception or two other acceptable methods of contraception, (e.g., intra-uterine device plus condom, spermicidal gel plus condom, diaphragm plus condom, etc.) from the time of randomization throughout the entire study.
   * Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   * Postmenopausal females must have had no menstrual bleeding for at least 1 year prior to inclusion in MYL-GAI-3001 study.
   * Female patients who report surgical sterilization must have had the procedure at least 6 months prior to inclusion to MYL-GAI-3001 study.
   * All female patients of childbearing potential, must have negative pregnancy test results at baseline (week 0) and at each clinic visit as per the SCHEDULE OF ACTIVITIES.
   * If female patients have male partners who have undergone vasectomy, the vasectomy must have occurred more than 6 months prior to inclusion in MYL-GAI-3001 study.

Exclusion Criteria:

1. History or presence of a medical condition or disease that in the Investigator's opinion would place the patient at an unacceptable risk from trial participation.
2. History of clinically significant (i.e., significant enough to alter the insulin dose requirement, as per the Investigator) acute bacterial, viral or fungal systemic infections in the 4 weeks prior to inclusion / randomization (recorded while collecting patient history) in to the MYL-1501D-3003 extension study
3. Patients scheduled to receive another investigational drug during the extension study period
4. Any major elective surgery requiring hospitalization planned during the extension study period.
5. Moderate insulin resistance, defined as requiring insulin (Basal + Prandial) of ≥1.5 U/kg/day (Lantus® in U/kg/day or Mylan's insulin glargine in IU/kg/day).

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blevins, Principal Investigator — Texas Diabetes & Endocrinology
Locations (76):
- United States (39):
  - Mylan Investigator Site, Fresno, California
  - Mylan Investigator Site, Greenbrae, California
  - Mylan Investigator Site, La Jolla, California
  - Mylan Investigator Site, Northridge, California
  - Mylan Investigator Site, Tustin, California
  - Mylan Investigator Site, Fort Lauderdale, Florida
  - Mylan Investigator Site, New Port Richey, Florida
  - Mylan Investigator Site, Palm Harbor, Florida
  - Mylan Investigator Site, West Palm Beach, Florida
  - Mylan Investigator Site, Atlanta, Georgia
  - Mylan Investigator Site, Columbus, Georgia
  - Mylan Investigator Site, Idaho Falls, Idaho
  - Mylan Investigator Site, Crystal Lake, Illinois
  - Mylan Investigator Site, Springfield, Illinois
  - Mylan Investigator Site, Des Moines, Iowa
  - Mylan Investigator Site, Overland Park, Kansas
  - Mylan Investigator Site, Lexington, Kentucky
  - Mylan Investigator Site, Billings, Montana
  - Mylan Investigator Site, Omaha, Nebraska
  - Mylan Investigator Site, Albany, New York
  - Mylan Investigator Site, Staten Island, New York
  - Mylan Investigator Site, Syracuse, New York
  - Mylan Investigator Site, Asheville, North Carolina
  - Mylan Investigator Site, Burlington, North Carolina
  - Mylan Investigator Site, Greenville, North Carolina
  - Mylan Investigator Site, Morehead City, North Carolina
  - Mylan Investigator Site, Wilmington, North Carolina
  - Mylan Investigator Site, Cincinnati, Ohio
  - Mylan Investigator Site, Mentor, Ohio
  - Mylan Investigator Site, Chattanooga, Tennessee
  - Mylan Investigator Site, Austin, Texas
  - Mylan Investigator Site, Dallas, Texas
  - Mylan Investigator Site, San Antonio, Texas
  - Mylan Investigator Site, Ogden, Utah
  - Mylan Investigator Site, Salt Lake City, Utah
  - Mylan Investigator Site, Chesapeake, Virginia
  - Mylan Investigator Site, Renton, Washington
  - Mylan Investigator Site, Tacoma, Washington
  - Mylan Investigator Site, Vancouver, Washington
- Canada (5):
  - Mylan Investigator Site, Red Deer, Alberta
  - Mylan Investigator Site., Vancouver, British Columbia
  - Mylan Investigator Site, Winnipeg, Manitoba
  - Mylan Investigator Site, Laval, Quebec
  - Mylan Investigator Site, Montreal, Quebec
- Czechia (5):
  - Mylan Investigator Site, Brno-Bohunice
  - Mylan Investigator Site, České Budějovice
  - Mylan Investigator Site, Olomouc
  - Mylan Investigator Site, Pardubice
  - Mylan Investigator Site, Prague
- Estonia (3):
  - Mylan Investigator Site, Pärnu
  - Mylan Investigator Site, Tallinn
  - Mylan Investigator Site, Tartu
- Germany (4):
  - Mylan Investigator Site, Aschaffenburg, Bavaria
  - Mylan Investigator Site, Münster, North Rhine-Westphalia
  - Mylan Investigator Site, Hohenmölsen, Saxony-Anhalt
  - Mylan Investigator Site, Hamburg
- Hungary (5):
  - Mylan Investigator Site, Budapest
  - Mylan Investigator Site, Eger
  - Mylan Investigator Site, Létavértes
  - Mylan Investigator Site, Miskolc
  - Mylan Investigator Site, Szeged
- Latvia (5):
  - Mylan Investigator Site, Limbaži
  - Mylan Investigator Site, Ogre
  - Mylan Investigator Site, Riga
  - Mylan Investigator Site, Sigulda
  - Mylan Investigator Site, Talsi
- Slovakia (10):
  - Mylan Investigator Site, Bratislava
  - Mylan Investigator Site, Dolný Kubín
  - Mylan Investigator Site, Levice
  - Mylan Investigator Site, Ľubochňa
  - Mylan Investigator Site, Nové Zámky
  - Mylan Investigator Site, Prievidza
  - Mylan Investigator Site, Rimavská Sobota
  - Mylan Investigator Site, Štúrovo
  - Mylan Investigator Site, Trebišov
  - Mylan Investigator Site, Žilina

RESULTS

PARTICIPANT FLOW:
Groups:
- Mylan's Insulin Glargine Sequence: Patients will be administered either Mylan insulin glargine or Lantus® subcutaneously, once daily in combination with lispro and titrated based on blood glucose readings per standard of care for a total of thirty-six (36) weeks, split into three cycles of twelve (12) weeks each.
  Mylan's insulin glargine
- Lantus® Sequence: Patients will be administered either Mylan insulin glargine or Lantus® subcutaneously, once daily in combination with lispro and titrated based on blood glucose readings per standard of care for a total of thirty-six (36) weeks, split into three cycles of twelve (12) weeks each.
  Lantus®
Period: Baseline
Arm/Group | Mylan's Insulin Glargine Sequence | Lantus® Sequence
Started | 64 | 63
Completed | 64 | 63
Not Completed | 0 | 0
Period: Period 1
Arm/Group | Mylan's Insulin Glargine Sequence | Lantus® Sequence
Started | 64 | 63
Completed | 63 | 62
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | Mylan's Insulin Glargine Sequence | Lantus® Sequence
Started | 63 | 62
Completed | 62 | 58
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 4
Period: Period 3
Arm/Group | Mylan's Insulin Glargine Sequence | Lantus® Sequence
Started | 62 | 58
Completed | 61 | 58
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mylan's Insulin Glargine: Patients will be administered either Mylan insulin glargine or Lantus® subcutaneously, once daily in combination with lispro and titrated based on blood glucose readings per standard of care for a total of thirty-six (36) weeks, split into three cycles of twelve (12) weeks each.
  Mylan's insulin glargine
- Lantus®: Patients will be administered either Mylan insulin glargine or Lantus® subcutaneously, once daily in combination with lispro and titrated based on blood glucose readings per standard of care for a total of thirty-six (36) weeks, split into three cycles of twelve (12) weeks each.
  Lantus®
- Total: Total of all reporting groups
Arm/Group | Mylan's Insulin Glargine | Lantus® | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (11.43) | 43.2 (12.69) | 44.0 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 27 | 50
  Male | 41 | 36 | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 0 | 2
  Black | 2 | 2 | 4
  Hispanic | 1 | 0 | 1
  White | 59 | 61 | 120
Region of Enrollment [Number; unit: participants]
  Europe | 30 | 27 | 57
  North America | 34 | 36 | 70
Dosing Time [Number; unit: participants]
  Morning | 11 | 12 | 23
  Evening | 53 | 51 | 104
Baseline HIV Status [Number; unit: participants]
  Negative | 64 | 62 | 126
  Positive | 0 | 1 | 1
Hepatitis B surface antigen (HBsAg) [Number; unit: participants]
  Negative | 64 | 63 | 127
  Positive | 0 | 0 | 0
Baseline hepatitis C antibody (HCVAb) [Number; unit: participants]
  Low positive | 0 | 1 | 1
  Negative | 64 | 62 | 126
Weight [Mean (Standard Deviation); unit: kilograms] | 80.712 (16.5393) | 82.415 (15.2942) | 81.557 (15.8936)
Height [Mean (Standard Deviation); unit: centimeters] | 173.299 (9.9451) | 174.092 (8.5502) | 173.692 (9.2511)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.744 (4.1795) | 27.134 (4.4084) | 26.937 (4.2820)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 21.369 (12.8879) | 20.212 (8.9657) | 20.801 (11.1013)
Baseline fasting plasma glucose [Mean (Standard Deviation); unit: mmol/L] | 9.82 (3.455) | 9.51 (4.099) | 9.67 (3.779)
Baseline hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: %] | 7.64 (0.997) | 7.87 (0.913) | 7.75 (0.959)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (HbA1c) From Baseline
Time Frame: Baseline to 36 weeks
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 61 | 57
percent | -0.05 (0.032) | -0.06 (0.034)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
mmol/L | -0.56 (3.458) | 0.10 (4.521)

3. Secondary Outcome: Overall Average of Self-monitoring Blood Glucose (SMBG) Change From Baseline
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
mmol/L | -0.144 (1.2569) | -0.426 (1.1243)

4. Secondary Outcome: Change From Baseline Total Daily Insulin Dose
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: Units per kilogram
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
Units per kilogram | 0.0016 (0.09239) | 0.0023 (0.07712)

5. Secondary Outcome: Local and Systemic Allergic Reactions
Time Frame: Baseline to 40 weeks
Measure: Number; unit: participants
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
participants
  Local | 1 | 1
  Systemic | 1 | 0

6. Secondary Outcome: Hypoglycemic Rate
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: episodes/30 days
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
episodes/30 days | 0.627 (2.7180) | 0.410 (4.0911)

7. Secondary Outcome: Hypoglycemic Incidence
Time Frame: Baseline to 36 weeks
Measure: Number; unit: events
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
events | 58 | 57

8. Secondary Outcome: Change From Baseline in Total Insulin Antibodies - Mylan Insulin Glargine Assay
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: percent binding
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
percent binding | -2.098 (5.3826) | -2.474 (5.2505)

9. Secondary Outcome: Change From Baseline in Total Insulin Antibodies - Lantus Assay
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: percent binding
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
percent binding | -1.288 (4.9617) | -2.351 (5.374)

10. Secondary Outcome: Change From Baseline in Cross-Reactive Insulin Antibody - Mylan Insulin Glargine Assay
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: percent binding
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
percent binding | -2.051 (5.3697) | -2.252 (5.1904)

11. Secondary Outcome: Change From Baseline in Cross-Reactive Insulin Antibody - Lantus Assay
Time Frame: Baseline to 36 weeks
Measure: Mean (Standard Deviation); unit: percent binding
Arm/Group | Mylan's Insulin Glargine | Lantus®
Number analyzed (Participants) | 64 | 63
percent binding | -1.232 (4.8965) | -2.192 (5.1741)

ADVERSE EVENTS:
Time Frame: 40 weeks
Arm/Group | Mylan's Insulin Glargine Sequence | Lantus® Sequence
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/63
Serious Adverse Events (participants affected / at risk) | 2/64 | 5/63
Other Adverse Events (participants affected / at risk) | 41/64 | 42/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mylan's Insulin Glargine Sequence (N=64) | Lantus® Sequence (N=63)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mylan's Insulin Glargine Sequence (N=64) | Lantus® Sequence (N=63)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Seasonal allergy (Immune system disorders) | 3 (4) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 2 (2) | 0 (0)
Stress (Psychiatric disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 3 (3)
Influenza (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (8)
Sinusitis (Infections and infestations) | 2 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 5 (7)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa fungal (Infections and infestations) | 0 (0) | 1 (1)
Periodontis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-05-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT02666430/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT02666430/SAP_001.pdf